CLINICAL TRIAL: NCT01204710
Title: A Randomized Phase 2 Study of Human Anti-PDGFRα Monoclonal Antibody IMC-3G3 Plus Mitoxantrone Plus Prednisone or Mitoxantrone Plus Prednisone in Metastatic Castration-Refractory Prostate Cancer Following Disease Progression or Intolerance on Docetaxel-based Chemotherapy
Brief Title: A Study of Olaratumab (IMC-3G3) in Prostate Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 13938; I5B-IE-JGDD (Other: Eli Lilly and Company); CP15-0805 (Other: ImClone Systems); 2009-018015-11 (EudraCT Number)
Record Dates: First submitted 2010-09-16; First posted 2010-09-17 (Estimated); Results first posted 2018-11-02 (Actual); Last update posted 2019-09-20 (Actual); Status verified 2019-09

CONDITIONS: Prostate Cancer
Keywords: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — olaratumab; Mitoxantrone; Prednisone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Olaratumab + Mitoxantrone (Experimental): 1 cycle = 3 weeks (21 days)
  Interventions: Biological: Olaratumab; Drug: Mitoxantrone; Drug: Prednisone
- Mitoxantrone: Optional Olaratumab Monotherapy (Active Comparator): 1 cycle = 3 weeks (21 days)
  Participants who experience progressive disease (PD) have the option to receive olaratumab monotherapy treatment.
  Interventions: Drug: Mitoxantrone; Drug: Prednisone

INTERVENTIONS:
Biological: Olaratumab — 15 milligrams per kilogram (mg/kg) intravenous (IV) Days 1 and 8
  Other Names: IMC-3G3; LY3012207
  Arms: Olaratumab + Mitoxantrone
Drug: Mitoxantrone — Mitoxantrone 12 milligrams per square meter (mg/m²) IV Day 1
  Mitoxantrone is to be administered for up to 12 cycles (total cumulative dose of mitoxantrone is restricted to ≤144 mg/m²)
Drug: Prednisone — 5 mg orally (PO) twice daily (BID) on each day

SUMMARY:
This is a study evaluating the safety and efficacy of the monoclonal antibody olaratumab plus mitoxantrone plus prednisone compared to mitoxantrone plus prednisone in metastatic castration-refractory prostate cancer following disease progression or intolerance on docetaxel-based chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* histologically-confirmed adenocarcinoma of the prostate
* radiographic evidence of metastatic prostate cancer (Stage M1 or D2)
* has prostate cancer unresponsive or refractory to medical or surgical castration with a serum testosterone level of <50 nanograms per milliliter (ng/mL)
* has had disease progression or intolerance on docetaxel-based therapy
* prostate-specific antigen (PSA) ≥10 ng/mL
* all clinically significant toxic effects of prior surgery, radiotherapy, chemotherapy or hormonal therapy have resolved to ≤Grade 1, based on National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) version (v) 4.02
* participant has an Eastern Cooperative Oncology Group (ECOG) Performance Status 0-2
* adequate hematologic function
* adequate hepatic function
* adequate renal function
* urinary protein is ≤1 on dipstick or routine analysis
* life expectancy of more than 3 months
* fertile man with partners that are women of childbearing potential must use an adequate method of contraception during the study
* signed Informed Consent Document

Exclusion Criteria:

* concurrent active malignancy other than adequately treated nonmelanomatous skin cancer or other noninvasive or in situ neoplasms
* The participant has received more than 1 prior cytotoxic chemotherapy regimen for metastatic disease
* prior therapy with mitoxantrone for advanced prostate cancer
* The participant has a history of symptomatic congestive heart failure or has a pre study echocardiogram or multigated acquisition scan with left ventricular ejection fraction that is ≥10% below the lower limit of normal institutional range
* history of prior treatment with other agents that directly inhibit platelet-derived growth factor (PDGF) or platelet-derived growth factor receptors (PDGFR)
* known allergy to any of the treatment components: olaratumab, mitoxantrone, and/or prednisone
* radiotherapy within 21 days prior to first dose of olaratumab
* any investigational therapy within 30 days of randomization
* is receiving corticosteroids at a dose >5 mg prednisone PO BID or equivalent
* received prior strontium-89, rhenium-186, rhenium-188, or samarium-153 radionucleotide therapy and has either ongoing evidence of bone marrow dysfunction or poorly controlled bone pain
* has any ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, serious cardiac arrhythmia, psychiatric illness, active bleeding or pathological condition that carries a high risk of bleeding, or any other serious uncontrolled medical disorders
* known or suspected brain or leptomeningeal metastases
* known human immunodeficiency virus infection or acquired immunodeficiency syndrome-related illness

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 123 (Actual)
Dates: Start 2010-10; Primary Completion 2012-09 (Actual); Study Completion 2013-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (38):
- Belgium (3):
  - ImClone Investigational Site, Charleroi
  - ImClone Investigational Site, Edegem
  - ImClone Investigational Site, Liège
- Czechia (2):
  - ImClone Investigational Site, Olomouc
  - ImClone Investigational Site, Prague
- Germany (11):
  - ImClone Investigational Site, Aachen
  - ImClone Investigational Site, Augsburg
  - ImClone Investigational Site, Bonn
  - ImClone Investigational Site, Dresden
  - ImClone Investigational Site, Essen
  - ImClone Investigational Site, Frankfurt
  - ImClone Investigational Site, Freiburg im Breisgau
  - ImClone Investigational Site, Mainz
  - ImClone Investigational Site, Mannheim
  - ImClone Investigational Site, Münster
  - ImClone Investigational Site, Rostock
- Hungary (7):
  - ImClone Investigational Site, Budapest
  - ImClone Investigational Site, Debrecen
  - ImClone Investigational Site, Kecskemét
  - ImClone Investigational Site, Miskolc
  - ImClone Investigational Site, Nyíregyháza
  - ImClone Investigational Site, Pécs
  - ImClone Investigational Site, Szeged
- Italy (5):
  - ImClone Investigational Site, Meldola
  - ImClone Investigational Site, Milan
  - ImClone Investigational Site, Roma
  - ImClone Investigational Site, Rozzano
  - ImClone Investigational Site, Trento
- Poland (4):
  - ImClone Investigational Site, Krakow
  - ImClone Investigational Site, Lublin
  - ImClone Investigational Site, Poznan
  - ImClone Investigational Site, Warsaw
- Spain (6):
  - ImClone Investigational Site, Barcelona
  - ImClone Investigational Site, Madrid
  - ImClone Investigational Site, Palma de Mallorca
  - ImClone Investigational Site, Pamplona - Navarra
  - ImClone Investigational Site, Sabadell - Barcelona
  - ImClone Investigational Site, Valencia

IPD SHARING:
Plan to Share IPD: Yes
Anonymized individual patient level data will be provided in a secure access environment upon approval of a research proposal and a signed data sharing agreement.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data are available 6 months after the primary publication and approval of the indication studied in the US and EU, whichever is later. Data will be indefinitely available for requesting.
Access Criteria: A research proposal must be approved by an independent review panel and researchers must sign a data sharing agreement.
URL: https://vivli.org/

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A participant was considered to have completed the study if he or she experienced progressive disease (PD) or had died.
Groups:
- Olaratumab (IMC-3G3) + Mitoxantrone: 15 milligrams per kilogram (mg/kg) olaratumab was administered intravenously (IV) on Days 1 and 8 of each 21-day cycle, followed by 12 milligrams per square meter (mg/m²) mitoxantrone IV on Day 1 of each 21-day cycle with 5 milligrams (mg) prednisone orally (PO) twice daily (BID) on each day.
  Mitoxantrone was administered for up to 12 cycles (total cumulative dose of mitoxantrone was restricted to ≤144 mg/m²).
  After 12 cycles, participants continued to receive 15 mg/kg olaratumab IV on Days 1 and 8 of each 21-day cycle with 5 mg prednisone PO BID on each day until withdrawal criteria were met.
- Mitoxantrone: Optional Olaratumab Monotherapy: 12 mg/m² mitoxantrone was administered IV on Day 1 of each 21-day cycle with 5 mg prednisone PO BID on each day.
  Mitoxantrone was administered for up to 12 cycles (total cumulative dose of mitoxantrone is restricted to ≤144 mg/m²).
  Participants who experienced PD had the option to receive olaratumab monotherapy treatment. 15 mg/kg olaratumab was administered IV on Days 1 and 8 of each 21-day cycle with 5 mg prednisone PO BID on each day. Participants received treatment until withdrawal criteria were met.
Period: Randomization Treatment
Arm/Group | Olaratumab (IMC-3G3) + Mitoxantrone | Mitoxantrone: Optional Olaratumab Monotherapy
Started | 63 | 60
Received ≥1 Dose of Study Drug | 62 | 59
Completed | 49 | 47
Not Completed | 14 | 13
Not completed — Lost to Follow-up | 1 | 0
Not completed — Withdrawal by Subject | 6 | 5
Not completed — Physician Decision | 3 | 2
Not completed — Entry criteria not met | 0 | 1
Not completed — Adverse Event | 4 | 2
Not completed — Sponsor Decision | 0 | 1
Not completed — Worsening of General condition | 0 | 1
Not completed — Moved and Followed for Survival | 0 | 1
Period: Optional Olaratumab Monotherapy
Arm/Group | Olaratumab (IMC-3G3) + Mitoxantrone | Mitoxantrone: Optional Olaratumab Monotherapy
Started | 0 (Olaratumab follow-on treatment was optional for participants in mitoxantrone group only who had PD.) | 19 (Among 43 participants who experienced PD, 19 received olaratumab monotherapy.)
Completed | 0 | 16
Not Completed | 0 | 3
Not completed — Olaratumab Intolerance | 0 | 1
Not completed — Physician Decision | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Population: All randomized participants who received ≥1 dose of study drug.
Groups:
- Olaratumab + Mitoxantrone: 15 mg/kg olaratumab was administered IV on Days 1 and 8 of each 21-day cycle, followed by 12 mg/m² mitoxantrone IV on Day 1 of each 21-day cycle with 5 mg prednisone PO BID on each day.
  Mitoxantrone was administered for up to 12 cycles (total cumulative dose of mitoxantrone was restricted to ≤144 mg/m²).
  After 12 cycles, participants continued to receive 15 mg/kg olaratumab IV on Days 1 and 8 of each 21-day cycle with 5 mg prednisone PO BID on each day until withdrawal criteria were met.
- Total: Total of all reporting groups
Arm/Group | Olaratumab + Mitoxantrone | Mitoxantrone: Optional Olaratumab Monotherapy | Total
Number analyzed (Participants) | 62 | 59 | 121
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 20 | 15 | 35
  >=65 years | 42 | 44 | 86
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 62 | 59 | 121
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 3 | 5
  Not Hispanic or Latino | 60 | 56 | 116
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 62 | 58 | 120
  More than one race | 0 | 1 | 1
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  Hungary | 6 | 10 | 16
  Czechia | 5 | 2 | 7
  Spain | 17 | 12 | 29
  Poland | 11 | 6 | 17
  Belgium | 3 | 2 | 5
  Germany | 15 | 16 | 31
  Italy | 5 | 11 | 16

OUTCOME MEASURES:

1. Primary Outcome: Progression-Free Survival (PFS)
Description: PFS is measured from randomization to the earliest date of the following events: PD according to Response Evaluation Criteria In Solid Tumors (RECIST) criteria version (v) 1.1, is a ≥20% increase in the sum of diameter of the target lesions taking as reference the smallest sum on study and an absolute increase in the sum diameter of ≥5 millimeter (mm), the appearance of 1 or more new lesions and/or unequivocal progression of existing nontarget lesions, unequivocal evidence of progression by bone scan, clinical progression or death from any cause. For participants who had no documented PD or death or had started new anti-cancer therapy or were lost to follow-up, PFS was censored at their last tumor assessment.
Time Frame: Randomization to Measured PD or Death Due to Any Cause Up to 23 Months
Population: All randomized participants who received ≥1 dose of study drug. The number of participants censored was 10 for olaratumab + mitoxantrone group and 5 for mitoxantrone group.
Measure: Median (95% Confidence Interval); unit: months
Groups:
- Mitoxantrone: 12 mg/m² mitoxantrone was administered IV on Day 1 of each 21-day cycle with 5 mg prednisone PO BID on each day.
  Mitoxantrone was administered for up to 12 cycles (total cumulative dose of mitoxantrone is restricted to ≤144 mg/m²).
Arm/Group | Olaratumab + Mitoxantrone | Mitoxantrone
Number analyzed (Participants) | 62 | 59
months | 2.3 [2.2 to 2.8] | 2.4 [2.2 to 3.8]
Statistical Analysis 1: Comparison: Olaratumab + Mitoxantrone vs Mitoxantrone; Test type: Superiority or Other; p = 0.2201, Log Rank — Analysis was stratified by the randomization stratification factor: best overall response to prior docetaxel-based chemotherapy; Hazard Ratio (HR) = 1.29, 95% CI 2-sided [0.87 to 1.90] — Hazard ratio is expressed as IMC-3G3 + Mitoxantrone / Mitoxantrone and estimated from Cox model

2. Secondary Outcome: Overall Survival (OS)
Description: OS was defined as the time from the date of randomization to the date of death from any cause. If the participants were alive at the end of the follow-up period or were lost to follow-up, OS time was censored on the last date the participant was known to be alive.
Time Frame: Randomization to Death Due to Any Cause Up to 36 Months
Population: All randomized participants who received ≥1 dose of study drug. The number of participants censored was 12 for olaratumab + mitoxantrone group and 13 for mitoxantrone group.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Olaratumab + Mitoxantrone | Mitoxantrone
Number analyzed (Participants) | 62 | 59
months | 14.2 [12.2 to 16.0] | 12.8 [8.1 to 16.4]
Statistical Analysis 1: Comparison: Olaratumab + Mitoxantrone vs Mitoxantrone; Test type: Superiority or Other; p = 0.7291, Log Rank — [p-value comment as in outcome 1, analysis 1]; Hazard Ratio (HR) = 1.08, 95% CI 2-sided [0.72 to 1.61] — Hazard ratio is expressed as Olaratumab + Mitoxantrone / Mitoxantrone and estimated from Cox model

3. Secondary Outcome: Percentage of Participants Who Achieved a Best Overall Response of Complete Response (CR) or Partial Response (PR) [Objective Response Rate (ORR)]
Description: Best response is categorized using the RECIST v1.1 guidelines. CR is the disappearance of all non-nodal target lesions, with the short axes of any target lymph nodes reduced to <10 mm. PR is a ≥30% decrease in the sum of the diameters of target lesions (including the short axes of any target lymph nodes), taking as reference the pretreatment sum diameter. Percentage of participants = (number of participants who had CR or PR) / (number of participants treated) * 100.
Time Frame: Randomization to Objective PD or Death Up to 23 Months
Population: All randomized participants who received at least ≥1 dose of study drug and had measurable disease.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Olaratumab + Mitoxantrone | Mitoxantrone
Number analyzed (Participants) | 30 | 32
percentage of participants | 10.0 [3.5 to 25.6] | 3.1 [0.6 to 15.7]
Statistical Analysis 1: Comparison: Olaratumab + Mitoxantrone vs Mitoxantrone; Test type: Superiority or Other; p = 0.3465, Fisher Exact

4. Secondary Outcome: Percentage of Participants With a ≥50% Decrease in Prostate Specific Androgen (PSA) From Pretreatment to Any Time
Description: Decrease in PSA ≥50% from pretreatment required confirmation no less than 3 weeks after the initial suggestion of response and occurring prior to documentation of PD. Percentage of participants = (number of participants who had ≥50% decrease in PSA at any time) / (number of participants treated) * 100.
Time Frame: Pretreatment to PD Up to 23 Months
Population: All randomized participants who received ≥1 dose of study drug.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Olaratumab + Mitoxantrone | Mitoxantrone
Number analyzed (Participants) | 62 | 59
percentage of participants | 22.6 [14.0 to 34.4] | 18.6 [10.7 to 30.4]
Statistical Analysis 1: Comparison: Olaratumab + Mitoxantrone vs Mitoxantrone; Test type: Superiority or Other; p = 0.6571, Fisher Exact

5. Secondary Outcome: Percentage of Participants With a ≥30% Decrease in PSA From Pretreatment to Week 12
Description: Percentage of participants = (number of participants who had ≥30% decrease in PSA at Week 12) / (number of participants treated) * 100.
Time Frame: Pretreatment through Week 12
Population: All randomized participants who received ≥1 dose of study drug.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Olaratumab + Mitoxantrone | Mitoxantrone
Number analyzed (Participants) | 62 | 59
percentage of participants | 22.6 [14.0 to 34.4] | 16.9 [9.5 to 28.5]
Statistical Analysis 1: Comparison: Olaratumab + Mitoxantrone vs Mitoxantrone; Test type: Superiority or Other; p = 0.4986, Fisher Exact

6. Secondary Outcome: Summary Listing of Participants Reporting Treatment-Emergent Adverse Events (TEAE)
Description: Data presented are the number of participants who experienced serious adverse events (SAEs) and other nonserious adverse events (AEs). For participants in mitoxantrone group who had PD and chose optional IMC-3G3 follow-on treatment, the baseline was defined as the last assessment prior to the start of the olaratumab treatment. A summary of SAEs and other nonserious AEs, regardless of causality, is located in the Reported Adverse Events section.
Time Frame: From Start of Treatment Through Study Completion Up to 36 months
Population: All randomized participants who received at least 1 dose of study drug.
Measure: Number; unit: participants
Arm/Group | Olaratumab + Mitoxantrone | Mitoxantrone | Mitoxantrone: Optional Olaratumab Monotherapy
Number analyzed (Participants) | 62 | 59 | 19
participants
  SAEs | 26 | 21 | 6
  AEs | 52 | 51 | 15

7. Secondary Outcome: PFS Based on Baseline Circulating Tumor Cells (CTC) Counts
Description: High expression (HE) of CTC was defined as having CTC counts ≥5 cells/7.5 milliliter (mL) and low expression (LE) of CTC was defined as having CTC counts <5 cells/7.5 mL. PFS is measured from randomization to the earliest date of the following events: PD according to RECIST criteria v. 1.1, is a ≥20% increase in the sum diameter of the target lesions taking as reference the smallest sum on study and an absolute increase in the sum diameter of ≥5 mm, the appearance of 1 or more new lesions and/or unequivocal progression of existing nontarget lesions, unequivocal evidence of progression by bone scan, clinical progression or death from any cause.
Time Frame: Randomization to Measured PD or Death Due to Any Cause Up to 23 Months
Population: All randomized participants who had evaluable data for CTC counts at baseline. The CTC counts assessment across both arms, high and low expression, was pre-specified in the statistical analysis plan.
Measure: Median (95% Confidence Interval); unit: months
Groups:
- Olaratumab + Mitoxantrone (HE): Participants with CTC counts ≥5 cells/7.5 mL at baseline received 15 mg/kg olaratumab IV on Days 1 and 8 of each 21-day cycle, followed by 12 mg/m² mitoxantrone IV on Day 1 of each 21-day cycle with 5 mg prednisone PO BID on each day. Mitoxantrone was administered for up to 12 cycles (total cumulative dose of mitoxantrone was restricted to ≤144 mg/m²).
- Mitoxantrone (HE); Mitoxantrone (LE): 12 mg/m² mitoxantrone was administered IV on Day 1 of each 21-day cycle with 5 mg prednisone PO BID on each day.
  Mitoxantrone was administered for up to 12 cycles (total cumulative dose of mitoxantrone is restricted to ≤144 mg/m²).
- Olaratumab + Mitoxantrone (LE): Participants with CTC counts <5 cells/7.5 mL at baseline received 15 mg/kg olaratumab IV on Days 1 and 8 of each 21-day cycle, followed by 12 mg/m² mitoxantrone IV on Day 1 of each 21-day cycle with 5 mg prednisone PO BID on each day. Mitoxantrone was administered for up to 12 cycles (total cumulative dose of mitoxantrone was restricted to ≤144 mg/m²).
Arm/Group | Olaratumab + Mitoxantrone (HE) | Mitoxantrone (HE) | Olaratumab + Mitoxantrone (LE) | Mitoxantrone (LE)
Number analyzed (Participants) | 32 | 32 | 21 | 18
months | 2.32 [2.10 to 2.79] | 2.23 [2.10 to 2.40] | 2.38 [2.14 to 7.20] | 4.91 [2.40 to 11.73]

8. Secondary Outcome: OS Based on Baseline CTC Counts
Description: HE of CTC was defined as having CTC counts ≥5 cells/7.5 mL and LE of CTC was defined as having CTC counts <5 cells/7.5 mL. OS was defined as the time from the date of randomization to the date of death from any cause.
Time Frame: Randomization to Death Due to Any Cause Up to 36 Months
Population: as for outcome 7
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Olaratumab + Mitoxantrone (HE) | Mitoxantrone (HE) | Olaratumab + Mitoxantrone (LE) | Mitoxantrone (LE)
Number analyzed (Participants) | 32 | 32 | 21 | 18
months | 12.85 [7.10 to 15.18] | 8.10 [5.82 to 13.14] | 16.49 [9.13 to 28.12] | 23.00 [11.93 to NA] — The upper confidence interval for median OS is inestimable when the curve representing the upper confidence limits for the survivor function falls above the 0.5 line.

9. Secondary Outcome: Number of Participants With Negative Platelet-Derived Growth Factor Receptor Alpha (PDGFRα) Protein Expression by Immunohistochemistry (IHC)
Description: PDGFRα protein expression (pretreatment) by IHC was assessed in tumor cells, and was provided as a dichotomous variable with "positive" and "negative" expression. "Positive" corresponds to weak intensity membranous staining comprising greater than 30% of the tumor and/or moderate to strong intensity membranous staining comprising greater than 5% of the tumor. "Negative" corresponds to staining that does not meet these requirements.
Time Frame: Baseline
Population: All randomized participants who received at least 1 dose of study drug and provided tissue specimens from the initial diagnosis for PDGFRα protein expression analysis.
Measure: Number; unit: participants
Arm/Group | Olaratumab + Mitoxantrone | Mitoxantrone
Number analyzed (Participants) | 14 | 9
participants | 14 | 9

10. Other Pre Specified Outcome: Number of Participants Who Died During Study
Time Frame: From Start of Treatment through Study Completion up to 36 Months
Population: All randomized participants who received at least 1 dose of study drug.
Measure: Number; unit: participants
Arm/Group | Olaratumab + Mitoxantrone | Mitoxantrone | Mitoxantrone: Optional Olaratumab Monotherapy
Number analyzed (Participants) | 62 | 59 | 19
participants
  Due to PD | 43 | 27 | 12
  Due to AEs | 4 | 3 | 1
  Due to Other reasons | 3 | 2 | 1

11. Secondary Outcome: Percentage of Participants With Anti-Olaratumab Antibody Assessment (Immunogenicity)
Description: Participants with Treatment Emergent (TE) anti-olaratumab antibodies were participants with a 4-fold increase (2 dilutions) increase over a positive baseline antibody titer or for a negative baseline titer, a participant with an increase from the baseline to a level of 1:20.
Time Frame: From Start of Treatment up to 9 Months
Population: All randomized participants who received ≥1 dose of study drug and had evaluable baseline and evaluable post-baseline antibody data. The participants analyzed under Mitoxantrone are those in control arm receiving subsequent optional olaratumab monotherapy.
Measure: Number; unit: percent of participants
Arm/Group | Olaratumab + Mitoxantrone | Mitoxantrone
Number analyzed (Participants) | 52 | 11
percent of participants | 3.8 | 0

12. Secondary Outcome: Maximum Concentration (Cmax) of Olaratumab Cycles 1, 2 and 3
Time Frame: Day 1 of Cycles 1, 2 and 3, and Day 8 of Cycles 1 and 3 (21-day cycle)
Population: Zero participants were analyzed. An insufficient amount of samples were collected to obtain this measure.
Groups:
- Olaratumab+ Mitoxantrone: 15 mg/kg olaratumab was administered IV on Days 1 and 8 of each 21-day cycle, followed by 12 mg/m² mitoxantrone IV on Day 1 of each 21-day cycle with 5 mg prednisone PO BID on each day.
  Mitoxantrone was administered for up to 12 cycles (total cumulative dose of mitoxantrone was restricted to ≤144 mg/m²).
  After 12 cycles, participants continued to receive 15 mg/kg olaratumab IV on Days 1 and 8 of each 21-day cycle with 5 mg prednisone PO BID on each day until withdrawal criteria were met.
Arm/Group | Olaratumab+ Mitoxantrone
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Groups:
- Mitoxantrone: Optional Olaratumab Monotherapy: 12 mg/m² mitoxantrone was administered IV on Day 1 of each 21-day cycle with 5 mg prednisone PO BID on each day.
  Mitoxantrone was administered for up to 12 cycles (total cumulative dose of mitoxantrone is restricted to ≤144 mg/m²).
  Participants who experienced PD had the option to receive olaratumab monotherapy treatment.15 mg/kg olaratumab was administered IV on Days 1 and 8 of each 21-day cycle with 5 mg prednisone PO BID on each day. Participants received treatment until withdrawal criteria were met.
Arm/Group | Olaratumab + Mitoxantrone | Mitoxantrone | Mitoxantrone: Optional Olaratumab Monotherapy
Serious Adverse Events (participants affected / at risk) | 26/62 | 21/59 | 6/19
Other Adverse Events (participants affected / at risk) | 52/62 | 51/59 | 15/19
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Olaratumab + Mitoxantrone (N=62) | Mitoxantrone (N=59) | Mitoxantrone: Optional Olaratumab Monotherapy (N=19)
Agranulocytosis (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 5 (5) | 4 (4) | 1 (1)
Anaemia of malignant disease (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1) | 1 (2) | 0 (0)
Leukopenia (Blood and lymphatic system disorders) | 0 (0) | 2 (2) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 2 (4) | 3 (3) | 0 (0)
Pancytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 3 (3) | 0 (0) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 2 (2) | 1 (1) | 0 (0)
Atrial flutter (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Cardiac arrest (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Cardiac failure chronic (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Cardiac failure congestive (Cardiac disorders) | 1 (3) | 0 (0) | 0 (0)
Congestive cardiomyopathy (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Myocardial ischaemia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1)
Periodontitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Asthenia (General disorders) | 1 (2) | 0 (0) | 1 (1)
Fatigue (General disorders) | 0 (0) | 1 (1) | 0 (0)
General physical health deterioration (General disorders) | 1 (1) | 1 (1) | 0 (0)
Localised oedema (General disorders) | 0 (0) | 1 (1) | 0 (0)
Multi-organ failure (General disorders) | 1 (1) | 0 (0) | 0 (0)
Oedema peripheral (General disorders) | 0 (0) | 1 (1) | 0 (0)
Pain (General disorders) | 0 (0) | 1 (1) | 2 (2)
Anaphylactic reaction (Immune system disorders) | 2 (2) | 0 (0) | 0 (0)
Anaphylactic shock (Immune system disorders) | 1 (1) | 0 (0) | 1 (1)
Hypersensitivity (Immune system disorders) | 1 (1) | 0 (0) | 0 (0)
Bronchopneumonia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Erysipelas (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Gastroenteritis escherichia coli (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 3 (3) | 0 (0)
Rectal abscess (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Respiratory tract infection (Infections and infestations) | 2 (2) | 1 (1) | 0 (0)
Septic shock (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Urosepsis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Cystitis radiation (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Femur fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Incorrect dose administered (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Subdural haematoma (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
General physical condition abnormal (Investigations) | 0 (0) | 1 (1) | 1 (1)
Cachexia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 1 (1)
Bone pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 (3) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Cerebral haemorrhage (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Depressed level of consciousness (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Facial paresis (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Ischaemic stroke (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Muscle spasticity (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Paraparesis (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Paraplegia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Spinal cord compression (Nervous system disorders) | 1 (1) | 2 (2) | 0 (0)
Alcoholism (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Hydronephrosis (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Renal failure acute (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Urinary tract obstruction (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0) | 0 (0)
Pulmonary infarction (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Circulatory collapse (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 2 (2) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Olaratumab + Mitoxantrone (N=62) | Mitoxantrone (N=59) | Mitoxantrone: Optional Olaratumab Monotherapy (N=19)
Anaemia (Blood and lymphatic system disorders) | 17 (41) | 15 (33) | 3 (4)
Leukopenia (Blood and lymphatic system disorders) | 9 (25) | 8 (13) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 19 (44) | 11 (28) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 8 (19) | 6 (17) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 2 (2) | 4 (6) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 2 (2) | 2 (3) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 3 (4) | 0 (0)
Cheilitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 5 (6) | 11 (14) | 3 (4)
Diarrhoea (Gastrointestinal disorders) | 12 (15) | 7 (8) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 5 (6) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1)
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 15 (19) | 14 (19) | 2 (2)
Vomiting (Gastrointestinal disorders) | 5 (5) | 3 (3) | 1 (1)
Asthenia (General disorders) | 18 (39) | 13 (23) | 5 (5)
Fatigue (General disorders) | 11 (11) | 11 (13) | 3 (3)
Infusion related reaction (General disorders) | 1 (1) | 0 (0) | 2 (3)
Oedema peripheral (General disorders) | 6 (8) | 4 (4) | 1 (1)
Pyrexia (General disorders) | 4 (8) | 7 (7) | 1 (1)
Urinary tract infection (Infections and infestations) | 2 (2) | 1 (2) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 1 (1) | 1 (1) | 1 (1)
Ejection fraction decreased (Investigations) | 1 (1) | 3 (3) | 0 (0)
Gamma-glutamyltransferase increased (Investigations) | 2 (2) | 3 (5) | 0 (0)
Weight decreased (Investigations) | 2 (2) | 5 (6) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 11 (15) | 6 (10) | 3 (5)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 1 (1)
Hypovitaminosis (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Vitamin b12 deficiency (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 7 (7) | 3 (6) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 6 (8) | 7 (8) | 2 (2)
Bone pain (Musculoskeletal and connective tissue disorders) | 7 (10) | 5 (5) | 1 (1)
Flank pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (2) | 1 (1)
Muscle atrophy (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 4 (5) | 1 (1) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 4 (4) | 2 (2)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 7 (7) | 3 (4) | 0 (0)
Dizziness (Nervous system disorders) | 2 (3) | 3 (4) | 0 (0)
Dysgeusia (Nervous system disorders) | 2 (2) | 3 (4) | 0 (0)
Headache (Nervous system disorders) | 4 (6) | 5 (17) | 1 (1)
Paraesthesia (Nervous system disorders) | 1 (1) | 3 (3) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 2 (2) | 1 (1)
Depression (Psychiatric disorders) | 2 (2) | 1 (1) | 1 (1)
Haematuria (Renal and urinary disorders) | 2 (3) | 4 (5) | 0 (0)
Pollakiuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (2)
Urinary incontinence (Renal and urinary disorders) | 1 (1) | 4 (4) | 0 (0)
Urinary retention (Renal and urinary disorders) | 0 (0) | 0 (0) | 3 (4)
Pelvic pain (Reproductive system and breast disorders) | 3 (3) | 2 (2) | 2 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 6 (6) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 4 (5) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (2) | 1 (1)
Hypoaesthesia facial (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2) | 2 (2)
Skin disorder (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 5 (7) | 2 (6) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 3 (3) | 0 (0)
Thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
Efficacy analysis for the follow-on treatment is exploratory, therefore, efficacy analysis for follow-on treatment are not included in this clinical trial results.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Investigators agreed to delay independently publishing or disclosing data, findings or conclusions from the study except as part of a multi-center publication. Upon study publication or if draft publication is not produced within approximately 6 months of the final report of the study results, investigators may independently publish, subject to confidential information review/redaction by sponsor. Sponsor may request publication delay up to 90 days to seek patent protection.